CLINICAL TRIAL: NCT01939314
Title: A Prospective, Randomized, Double-Blind Study Comparing the Efficacy of Sphenopalatine Nerve Block by Localized Mucosal Application of an Anesthetic vs Placebo for the Emergency Department Management
Brief Title: Sphenopalatine Nerve Block for Headache Tx360
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jason Schaffer, Primary Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TX 360 HA -Schaffer; Tian Medical Inc. (Other: Tian Medical Inc)
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Headache; Migraine
Keywords: Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): Bupivicaine .03ml to each nare
  Interventions: Drug: Bupivacaine
- Normal Saline (Placebo Comparator): normal saline .03 ml to each nare
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — Bupivavaine Delivered by the Tx 360 Device to the Sphenopalatine Ganglion
  Arms: Bupivacaine
Drug: Placebo — Normal Saline Delivered by the Tx 360 Device to the Sphenopalatine Ganglion
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
The primary objective of this study is to evaluate the efficacy of sphenopalatine nerve block utilizing the Tx360 (device) to deliver an anesthetic agent (bupivacaine) and to assess the duration of the analgesia.

ELIGIBILITY:
Inclusion Criteria:

* are 18 - 65 years of age
* present to emergency department (ED) triage with chief complaint of crescendo-onset anterior/frontal headache (affecting frontal, temporal, orbital, maxillary, and mandible region)
* have a normal neurological exams

Exclusion Criteria:

* are less than 18 years old or greater than 65
* have any focal neurological dysfunction signs or symptoms
* have a posterior/occipital/cervicogenic source predominance of headache
* are febrile (oral temperature 37.7 C or 100 F) or signs of acute or chronic sinusitis, such as congestion, has been present more than 10 days, there is a high fever, the nasal mucus is an abnormal color, or complains of face pain or headaches
* have self treated with pain medication or anti-emetic 4 hours prior to arrival
* have a history of peripheral vascular disease, cancer, or HIV infection
* are known to be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason T Schaffer, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 165 Patients Identified
Pre-assignment Details: 93 Patients Enrolled 47 Patients Excluded 25 Patients Declined
Groups:
- Bupivacaine: Bupivicaine .03ml to each nare
  Bupivacaine: intervention
- Normal Saline: normal saline .03 ml to each nare
  Placebo: Placebo
Period: Overall Study
Arm/Group | Bupivacaine | Normal Saline
Started | 45 | 48
15 Minute Endpoint | 41 | 46
24 Hour Endpoint | 36 | 40
Completed | 36 | 40
Not Completed | 9 | 8
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Bupivacaine: Bupivacaine delivered by the Tx 360 device to the sphenopalatine ganglion bilaterally
- Normal Saline: Normal Saline delivered by the Tx 360 device to the sphenopalatine ganglion bilaterally
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Normal Saline | Total
Number analyzed (Participants) | 41 | 46 | 87
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [23 to 44] | 41 [29.25 to 51] | 39 [28.5 to 47.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 10 | 13 | 23
Median Baseline Headache Score [Median (Inter-Quartile Range); unit: units on a scale] — 0mm (No Pain) to 100mm (Maximum Pain) on 100mm Visual Analog Scale
  units on a scale | 80 [66 to 93] | 79 [64 to 91.75] | 79 [64.5 to 92.5]
Median Baseline Nausea Score [Median (Inter-Quartile Range); unit: units on a scale] — 0mm (No Nausea) to 100mm (Maximum Nausea) on 100mm Visual Analog Scale
  units on a scale | 29 [0 to 48] | 0 [0 to 45.5] | 20 [0 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported a 50% or Greater Reduction in Pain at 15 Minutes as Measured on the 100mm Visual Analog Scale
Time Frame: 15 minutes from dose
Measure: Number; unit: percentage of participants
Groups:
- Normal Saline: Normal Saline .03ml to each nare
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 41 | 46
percentage of participants | 48.8 | 41.3
Statistical Analysis 1: Comparison: Bupivacaine vs Normal Saline; Test type: Superiority or Other; Risk Difference (RD) = 7.5, 95% CI 2-sided [-13.0 to 27.1]

2. Secondary Outcome: Categorical Pain Relief
Description: Categorical Pain Relief at 15 minutes. Participants were asked to categorize their pain relief at 15 minutes as "No", "Little", "Some", "A Lot" or "Complete". The table displays the number of participants who identified their pain relief in the categories provided.
Time Frame: 15 minutes from dose
Measure: Number; unit: participants
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 41 | 46
participants
  No Pain Relief | 13 | 13
  A Little Pain Relief | 6 | 9
  Some Pain Relief | 3 | 8
  A Lot of Pain Relief | 11 | 10
  Complete Pain Relief | 8 | 6

3. Secondary Outcome: Headache Free at 24 Hours
Description: The percentage of patients that were headache free at 24 hours by follow-up phone conversation.
Time Frame: 24 hours
Measure: Number; unit: percentage of participants
Arm/Group | Bupivacaine | Normal Saline
Number analyzed (Participants) | 36 | 40
percentage of participants | 72.2 | 47.5
Statistical Analysis 1: Comparison: Bupivacaine vs Normal Saline; Test type: Superiority or Other; Risk Difference (RD) = 24.7, 95% CI 2-sided [2.6 to 43.6]

ADVERSE EVENTS:
Time Frame: 24 Hours
Description: At 24 hour phone contact we assesses for any nasopharyngeal symptoms, ongoing headache or nausea, or other adverse events.
Arm/Group | Bupivacaine | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/46
Other Adverse Events (participants affected / at risk) | 5/41 | 3/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine (N=41) | Normal Saline (N=46)
Nasal Congestion (General disorders) | 2 | 1
Sore Throat (General disorders) | 1 | 0
Minor Epistaxis (Injury, poisoning and procedural complications) | 0 | 2
Hoarseness (General disorders) | 1 | 0
Nasal Dryness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No